CLINICAL TRIAL: NCT04577339
Title: The BCAE Study: Best Care for Abdominal Emergencies
Brief Title: The Best Care for Abdominal Emergencies Study
Acronym: BCAE
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/72
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2023-04

CONDITIONS: Acute Abdomen; Bowel Obstruction; Bowel; Ischemic, Acute; Bowel Perforated; Peritonitis
Keywords: peritonitis; acute abdomen; laparotomy; laparoscopy; interventional radiology; risk assessment; care guidelines
MeSH Terms: conditions — Abdomen, Acute; Intestinal Obstruction; Ischemia; Intestinal Perforation; Peritonitis | interventions — Laparotomy; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with acute abdominal conditions: All adult patients >=16years of age on all general adult wards (excluding maternity) between 2013 and 2020 with the following inclusion and exclusion criteria:
  Inclusion criteria:
  * Must have an acute intestinal condition, based on their ICD-10 codes and OPSC-4 codes
  * Must be >= 16 years of age at the time of admission
  * Have at least one full set of vital signs recorded on the day of admission
  * Have at least one full set of routine blood tests recorded on the day of admission
  Exclusion criteria:
  * Maternity admissions during/after pregnancy
  * Patients admitted or undergoing abdominal surgery for a second time or more
  Interventions: Procedure: Laparotomy or laparoscopy

INTERVENTIONS:
Procedure: Laparotomy or laparoscopy — Laparotomy is the opening of the abdominal cavity usually through a midline incision.
  Laparoscopy is using minimal access keyhole surgery to perform the surgery instead of laparotomy Interventional radiology is the use of imaging to perform a procedure on the abdomen without surgery, for example, using ultrasound to guide a needle to drain an abscess Best supportive care is usually end-of-life care concentration on relieving symptoms rather than treating the cause.
  Other Names: Interventional radiology; Best supportive care

SUMMARY:
This is a single-centre retrospective cohort study utilising electronic hospital records.

The aim of this study is to improve care for all patients with an intestinal emergency, irrespective of whether they have surgery or not. Data will be derived from electronic patient records collected as part of routine clinical patient care on all general adult wards (excluding maternity) between 2013 and 2020. The investigators will then identify patients who had an emergency laparotomy, and those who had a laparoscopic procedure. The investigators aim to identify 2 further groups where treatment is non-surgical (but could be medical or interventional radiology) or where treatment is considered futile, suggesting that an early focus on end of life care might be appropriate. The primary objective is to provide mortality rates for different treatment options, and analysis of short- and long-term outcomes. The secondary endpoints are to define patient sub-groups with similar health characteristics based on clinical data and an established risk index and to use statistical analysis to predict the risk of death for each patient group and treatment option, which will allow the investigators to identify the best care pathways for each cluster.

DETAILED DESCRIPTION:
Abdominal emergencies are common, involving perforation, obstruction or ischaemia of the bowel, often needing life-saving emergency surgery, with a large incision to access the abdominal cavity called "laparotomy". This procedure is high risk with 10% mortality rate. 30,000 emergency laparotomies are performed each year in England and Wales. Since 2013, the National Emergency Laparotomy Audit (NELA) has set standards of care and monitored outcomes for emergency laparotomy, which has reduced mortality from 11.8 to 9.5%. However, patients who do NOT have a laparotomy are not well characterised and do not receive the prioritised care patients having surgery do, even though their condition is no less severe. Initial research has shown a surprisingly large group of patients (32%) with an intestinal emergency do not have surgery and have 30-day mortality of 63%. There are three additional groups of patients admitted with abdominal emergencies: patients having keyhole surgery or interventional radiological procedures, and patients for whom any treatment would be futile and would benefit most from an end of life care pathway. Clearly further work is needed to investigate the management of ALL patients with intestinal emergency, to optimise care for each group of patients.The aim of this study is to improve care for all patients with an intestinal emergency, irrespective of whether they have surgery or not.

AIM:

This is a single-centre retrospective cohort study utilising electronic hospital records.

STUDY DESIGN:

Data will be derived from electronic patient records collected as part of routine clinical patient care on all general adult wards (excluding maternity) between 2013 and 2020.

Inclusion criteria:

* Must have an acute intestinal condition, based on their ICD-10 codes and OPSC-4 codes
* Must be >= 16 years of age at the time of admission
* Have at least one full set of vital signs recorded on the day of admission
* Have at least one full set of routine blood tests recorded on the day of admission

Exclusion criteria:

* Maternity admissions during/after pregnancy
* Patients admitted or undergoing abdominal surgery for a second time or more Using OPCS-4 codes from PAS and TheatreManTM and NELA data, the investigators will then identify patients who had an emergency laparotomy, and those who had a laparoscopic procedure. We aim to identify a further group where treatment is futile, suggesting that an early focus on end of life care might be appropriate.

The investigators have estimated that we will have about 2,500 patients who fulfil the inclusion criteria in this period. Patient outcomes will be analysed from up to one year following their admission for acute abdomen.

PRIMARY OBJECTIVE:

To provide mortality rates for different treatment options, and analysis of short- and long-term outcomes.

SECONDARY OBJECTIVE:

To define patient sub-groups with similar health characteristics based on clinical data and an established risk index, and to use statistical analysis to predict the risk of death for each patient group and treatment option, which will allow us to identify the best care pathways for each cluster.

PRIMARY ENDPOINT:

The mortality risk for each treatment group

SECONDARY ENDPOINT:

The risk of other outcomes and long-term complications and association between patient factors and these outcomes

ELIGIBILITY:
Inclusion Criteria:

All acute general surgical adult patients admitted between 2013 and 2020 with all of the conditions below:

* Must have an acute intestinal condition, based on their ICD-10 codes and OPSC-4 codes
* Must be >= 16 years of age at the time of admission
* Have at least one full set of vital signs recorded on the day of admission
* Have at least one full set of routine blood tests recorded on the day of admission

Exclusion Criteria:

* Maternity admissions during/after pregnancy
* Patients admitted or undergoing abdominal surgery for a second time or more

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All acute general surgical adult patients admitted between 2013 and 2020 presenting with an acute abdomen due to an underlying acute intestinal condition to a single centre (an Acute NHS Hospital in UK).
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Mortality rates of different interventions | 2013-2020
  Provide mortality rates for different treatment options, and analysis of short- and long-term outcomes.

SECONDARY OUTCOMES:
Define patient sub-groups with similar health characteristics | 2013-2020
  Define patient sub-groups with similar health characteristics based on clinical data and an established risk index.
  option, which will allow us to identify the best care pathways for each cluster.
Predict the risk of death for each patient group | 2013-2020
  Use statistical analysis to predict the risk of death for each patient group and treatment option, which will allow us to identify the best care pathways for each cluster.

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals University NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised patient data will be shared with our research partners in the Faculty of Health Modelling, University of Portsmouth
Supporting Information: Study Protocol, SAP
Time Frame: December 1st 2021 and for up to 2 years
Access Criteria: Only fully anonymised data will leave the study site in strict accordance with GDPR and DPA.

REFERENCES:
- See also: The BCAE Study website — https://stoh932714.wixsite.com/website-2

DOCUMENTS (1):
  • Study Protocol (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT04577339/Prot_000.pdf